CLINICAL TRIAL: NCT05948176
Title: Motor Development of Normal Children in Urban Versus Rural Regions
Brief Title: Motor Development of Normal Children
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadeer Abdallah Abdel Khalik, Physical therapist, Cairo University
Other Study IDs: P.T.REC/012/004138
Record Dates: First submitted 2023-07-08; First posted 2023-07-17 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Motor Development
Keywords: Motor development; Pre-school children; Urban and Rural areas; BOT2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Urban group1: 150 boys
  Interventions: Other: The Bruininks-Oseretsky Test of Motor Proficiency, Second Edition
- Urban group2: 150 girls
  Interventions: Other: The Bruininks-Oseretsky Test of Motor Proficiency, Second Edition
- Rural group 3: 150 boys
  Interventions: Other: The Bruininks-Oseretsky Test of Motor Proficiency, Second Edition
- Rural group 4: 150 girls
  Interventions: Other: The Bruininks-Oseretsky Test of Motor Proficiency, Second Edition

INTERVENTIONS:
Other: The Bruininks-Oseretsky Test of Motor Proficiency, Second Edition — It is a standardized measure of fine and gross motor skills in children and youth aged 4-21 years

SUMMARY:
The goal of this type of study: observational study is to compare motor development between urban and rural regions in pre-school age children. The main questions it aims to answer are:

* Is there difference in gross motor development of normal children aged from four to six years between urban and rural areas?
* Is there difference in fine motor development of normal children aged from four to six years between urban and rural areas?

Participants will be asked to perform tasks of bruininks-oseretsky test of motor proficiency, second edition.

Researchers will compare urban group and rural group to see if there is any difference in motor development.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-school normal children of both sexes.
2. Age will range from four to six years.

Exclusion Criteria:

1. Past history of any diseases or injuries during pregnancy and labor period.
2. History of cardiac or respiratory diseases.
3. Neurological disorders.
4. Visual or auditory defects.
5. Congenital or acquired deformities

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects will be selected from kindergartens.Subjects will be divided into two subgroups according to region . Each subgroup will be divided into two subgroups according to age and will contain 150 children.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Assessing motor development by Bruininks-Oseretsky Test of Motor Proficiency-2 (BOT-2) | Baseline
  BOT-2 is a norm-referenced standardized measure of fine and gross motor skills in children and youth aged 4-21 years.It consists of 53 items and is typically completed in 45-60 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Eman IB EL-Hadidy, Professor, Study Chair — Cairo University; Samia AB Abdel Rahman, Professor, Study Director — Cairo University; Hadeer AA Abdel El-Khalik, Masters, Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - Faculty of physical therapy,Cairo university, Cairo, Cairo Governorate
  - Schools, Cairo

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Results will be published by the investigators in academic journals.Sharing of generated study data will be carried out in several different ways.We plan to make our results available to researchers and potential collaborators

REFERENCES:
- [Background] Al-Thumali F (2016): Assessment of Motor Proficiency Levels in Children in Saudi Arabia. Theses and Dissertations. School of Education and Professional Studies, Griffith University, 7 (2):3-12.
- [Background] Balasundaram P, Avulakunta ID. Human Growth and Development. 2023 Mar 8. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK567767/ PMID 33620844
- [Background] Bellman M, Byrne O, Sege R. Developmental assessment of children. BMJ. 2013 Jan 15;346:e8687. doi: 10.1136/bmj.e8687. No abstract available. PMID 23321410
- [Background] Beltre G, Mendez MD. Child Development. 2023 Nov 13. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK564386/ PMID 33232056
- [Background] Bruininks R and Bruininks B (2005): Bruininks-oseretsky test of motor proficiency second edition manual. Minneapolis, MN: Pearson Assessments
- [Background] Bruininks RH and Bruinicks BD (2005): Bruininks-Oseretsky test of motor proficiency, second edition (BOT-2). Minneapolis, MN: Pearson. Accessed 21 May 2022
- [Background] Burkett T (2018): Norm-Referenced Testing and Criterion-Referenced Testing. In: Liontas JI (ed.): The TESOL Encyclopedia of English Language Teaching. John Wiley & Sons, Inc. pp:1-5.
- [Background] Cairney J, Hay J, Veldhuizen S, Missiuna C, Faught BE. Comparing probable case identification of developmental coordination disorder using the short form of the Bruininks-Oseretsky Test of Motor Proficiency and the Movement ABC. Child Care Health Dev. 2009 May;35(3):402-8. doi: 10.1111/j.1365-2214.2009.00957.x. PMID 19397603
- [Background] Case-smith J (2015): Development of childhood occupations. In: Case-smith j. and O'Brien J. (eds.): Occupational Therapy for Children and Adolescents. 7th edition. St Louis, MI: Elsevier Mosby. pp:67-69.
- [Background] Choo YY, Agarwal P, How CH, Yeleswarapu SP. Developmental delay: identification and management at primary care level. Singapore Med J. 2019 Mar;60(3):119-123. doi: 10.11622/smedj.2019025. PMID 30997518
- [Background] Cools W, Martelaer KD, Samaey C, Andries C. Movement skill assessment of typically developing preschool children: a review of seven movement skill assessment tools. J Sports Sci Med. 2009 Jun 1;8(2):154-68. PMID 24149522
- [Background] Cowden J and Torrey C (2007): Motor Development and Movement Activities for Preschoolers and Infants With Delays: A Multisensory Approach for Professionals and Families. 2nd edition. Charles C. Thomas Pub Ltd. pp:3-17.
- [Background] Croce RV, Horvat M, McCarthy E. Reliability and concurrent validity of the movement assessment battery for children. Percept Mot Skills. 2001 Aug;93(1):275-80. doi: 10.2466/pms.2001.93.1.275. PMID 11693695
- [Background] Deitz JC, Kartin D, Kopp K. Review of the Bruininks-Oseretsky Test of Motor Proficiency, Second Edition (BOT-2). Phys Occup Ther Pediatr. 2007;27(4):87-102. PMID 18032151
- [Background] Ferreira L, Godinez I, Gabbard C, Vieira JLL, Cacola P. Motor development in school-age children is associated with the home environment including socioeconomic status. Child Care Health Dev. 2018 Nov;44(6):801-806. doi: 10.1111/cch.12606. Epub 2018 Jul 31. PMID 30066336
- [Background] Ferreira L, Vieira J, Rocha F, Silva P, Cheuczuk F, Caçola P and Chaves R(2020): Percentile curves for Brazilian children evaluated with the Bruininks-Oseretsky Test of Motor Proficiency, 2nd edition. Revista Brasileira de Cineantropometria & Desempenho Humano, 22:e65027.
- [Background] Flensborg-Madsen T, Gronkjaer M, Mortensen EL. Predictors of early life milestones: Results from the Copenhagen Perinatal Cohort. BMC Pediatr. 2019 Nov 9;19(1):420. doi: 10.1186/s12887-019-1778-y. PMID 31703689
- [Background] Fraietta L (2018): Standardized assessment tools commonly used in adapted physical education. Theses and Dissertations. Master of Science in Exercise and Sport Science-Physical Education Teaching, Adapted Physical Education Concentration, University of Wisconsin-La Crosse: 126
- [Background] Gharaei E, Shojaei M and Daneshfar A (2019): The validity and reliability of the Bruininks-Oseretsky Test of Motor Proficiency, second edition brief form in preschool children. Annals of Applied Sport Science, 7(2):3-12.
- [Background] Haibach-Beach P, Reidn G and Collier D (2011): Motor learning and development. 1st edition. Champaign, IL: Human Kinetics
- [Background] Haywood KM and Getchell N (2020): Introduction to motor development. In: Andrew L, Christrine M, Anne E and Patricia L (Eds): Life Span Motor Development. 7th edition. Champaign, IL: Human Kinetics. pp:4-5.
- [Background] Jirovec J, Musalek M, Mess F. Test of Motor Proficiency Second Edition (BOT-2): Compatibility of the Complete and Short Form and Its Usefulness for Middle-Age School Children. Front Pediatr. 2019 Apr 18;7:153. doi: 10.3389/fped.2019.00153. eCollection 2019. PMID 31065548
- [Background] Keenan T, Evan S, and Crowley K (2016): The principles of developmental psychology. In: Block L (ed.): An Introduction to Child Development. 3rd edition. London: SAGE Publications Ltd. pp:8-9.
- [Background] Lane H, Brown T. Convergent validity of two motor skill tests used to assess school-age children. Scand J Occup Ther. 2015 May;22(3):161-72. doi: 10.3109/11038128.2014.969308. Epub 2014 Oct 20. PMID 25328127
- [Background] Lipkin PH, Okamoto J; Council on Children with Disabilities; Council on School Health. The Individuals With Disabilities Education Act (IDEA) for Children With Special Educational Needs. Pediatrics. 2015 Dec;136(6):e1650-62. doi: 10.1542/peds.2015-3409. PMID 26620061
- [Background] Lister C and Baard M (2020): Effects of integrated movement programme on motor proficiency, visual-motor integration and scholastic achievement of Grade 1 learners in Nelson Mandela Bay, South Africa. African Journal for Physical Activity and Health Sciences, 26(1): 41-57
- [Background] Matheia M and Estabillo JA (2018): Assessment of fine and gross motor skills in children. In: Matson JL (ed.): Handbook of Childhood Psychopathology and Developmental Disabilities Assessment. Springer. pp:467-484.
- [Background] McBrien JL, Stewart J, Ezati BA (2016): Positive youth development in war-affected children in Uganda. Contemporary Journal of African Studies,4(1):29-56.
- [Background] McCarty M, Clifton R and Collard R (2001): The beginnings of tool use by infants and toddlers. Infancy, 2(2): 233-256
- [Background] Misirliyan SS and Huynh AP (2021): Development milestones. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing. Available from: https://www.ncbi.nlm.nih.gov/books/NBK557518/
- [Background] Noordin H, Suppiah P, Azmi A, Joummy A, Ching P and Isahak N (2019): Gross motor development among 7-9 years old children in Sabah. International Journal of Physiology, Nutrition and Physical Education, 4(1): 501-504.
- [Background] Pajek SV. Impact of the COVID-19 Pandemic on the Motor Development of Schoolchildren in Rural and Urban Environments. Biomed Res Int. 2022 May 17;2022:8937693. doi: 10.1155/2022/8937693. eCollection 2022. PMID 35607301
- [Background] Payne V and Isaacs L (2011): Human motor development: A lifespan approach. 8th edition. NewYork: McGraw Hill.
- [Background] Phillips D, Hennermann JB, Tylki-Szymanska A, Borgwardt L, Gil-Campos M, Guffon N, Amraoui Y, Geraci S, Ardigo D, Cattaneo F, Lund AM. Use of the Bruininks-Oseretsky test of motor proficiency (BOT-2) to assess efficacy of velmanase alfa as enzyme therapy for alpha-mannosidosis. Mol Genet Metab Rep. 2020 Apr 8;23:100586. doi: 10.1016/j.ymgmr.2020.100586. eCollection 2020 Jun. PMID 32292699
- [Background] Radanovic D, Dordevic D, Stankovic M, Pekas D, Bogataj S, Trajkovic N. Test of Motor Proficiency Second Edition (BOT-2) Short Form: A Systematic Review of Studies Conducted in Healthy Children. Children (Basel). 2021 Sep 9;8(9):787. doi: 10.3390/children8090787. PMID 34572219
- [Background] Richardson P (2015): Use of standardized tests in pediatric practice. In: Case-smith J and O'Brien J. (eds.): Occupational Therapy for Children and Adolescents. 7th edition. St Louis, MI: Elsevier Mosby. pp:163-189
- [Background] Ryan RM, Deci EL. Intrinsic and Extrinsic Motivations: Classic Definitions and New Directions. Contemp Educ Psychol. 2000 Jan;25(1):54-67. doi: 10.1006/ceps.1999.1020. PMID 10620381
- [Background] Scharf RJ, Scharf GJ, Stroustrup A. Developmental Milestones. Pediatr Rev. 2016 Jan;37(1):25-37; quiz 38, 47. doi: 10.1542/pir.2014-0103. PMID 26729779
- [Background] Schulz J, Henderson SE, Sugden DA, Barnett AL. Structural validity of the Movement ABC-2 test: factor structure comparisons across three age groups. Res Dev Disabil. 2011 Jul-Aug;32(4):1361-9. doi: 10.1016/j.ridd.2011.01.032. Epub 2011 Feb 16. PMID 21330102
- [Background] Sharma A. Developmental examination: birth to 5 years. Arch Dis Child Educ Pract Ed. 2011 Oct;96(5):162-75. doi: 10.1136/adc.2009.175901. Epub 2011 Mar 13. PMID 21402576
- [Background] de Souza JM, Verissimo Mde L. Child development: analysis of a new concept. Rev Lat Am Enfermagem. 2015 Nov-Dec;23(6):1097-104. doi: 10.1590/0104-1169.0462.2654. PMID 26626001
- [Background] Spencer JP, Clearfield M, Corbetta D, Ulrich B, Buchanan P, Schoner G. Moving toward a grand theory of development: in memory of Esther Thelen. Child Dev. 2006 Nov-Dec;77(6):1521-38. doi: 10.1111/j.1467-8624.2006.00955.x. PMID 17107442
- [Background] Tamplain P, Webster EK, Brian A and Valentini NC (2020): Assessment of motor development in childhood: Contemporary issues, considerations, and future directions. Journal of Motor Learning and Development, 8(2):391-409
- [Background] Thelen E, Corbetta D, Spencer JP. Development of reaching during the first year: role of movement speed. J Exp Psychol Hum Percept Perform. 1996 Oct;22(5):1059-76. doi: 10.1037//0096-1523.22.5.1059. PMID 8865616
- [Background] Thelen E, Corbetta D, Kamm K, Spencer JP, Schneider K, Zernicke RF. The transition to reaching: mapping intention and intrinsic dynamics. Child Dev. 1993 Aug;64(4):1058-98. PMID 8404257
- [Background] Wang HY, Long IM, Liu MF. Relationships between task-oriented postural control and motor ability in children and adolescents with Down syndrome. Res Dev Disabil. 2012 Nov-Dec;33(6):1792-8. doi: 10.1016/j.ridd.2012.05.002. Epub 2012 Jun 13. PMID 22699252
- [Background] Wuang YP, Su CY. Reliability and responsiveness of the Bruininks-Oseretsky Test of Motor Proficiency-Second Edition in children with intellectual disability. Res Dev Disabil. 2009 Sep-Oct;30(5):847-55. doi: 10.1016/j.ridd.2008.12.002. Epub 2009 Jan 31. PMID 19181480
- [Background] Wuang YP, Su CY, Huang MH. Psychometric comparisons of three measures for assessing motor functions in preschoolers with intellectual disabilities. J Intellect Disabil Res. 2012 Jun;56(6):567-78. doi: 10.1111/j.1365-2788.2011.01491.x. Epub 2011 Oct 12. PMID 21988314